CLINICAL TRIAL: NCT01827111
Title: Phase II Study of Abraxane Plus Ipilimumab in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1157; NCI-2014-01238 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic Melanoma; Advanced stage IV melanoma; Unresectable stage III mucosal melanoma; Cutaneous melanoma; Progression-free survival; (PFS); ABI-007; Nab-paclitaxel; Paclitaxel; Abraxane; Ipilimumab; Yervoy; BMS-734016; MDX010
MeSH Terms: conditions — Melanoma | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Paclitaxel; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABI-007 + Ipilimumab (Experimental): Starting dose of ABI-007 is 150 mg/m2 administered by vein on days 1, 8, 15 every 28 days. Ipilimumab 3 mg/kg by vein over 90 minutes on day 1. Ipilimumab dose repeated every 21 days for a total of 4 doses. Every 2 months for 6 months, then every 3 months for up to 2 years, participant contacted by telephone. Each call should last about 5 minutes.
  Interventions: Drug: ABI-007; Drug: Ipilimumab; Behavioral: Phone Call

INTERVENTIONS:
Drug: ABI-007 — Starting dose of ABI-007 is 150 mg/m2 administered by vein on days 1, 8, 15 every 28 days. The cycle length for ABI-007 is 28 days.
  Other Names: Nab-paclitaxel; Paclitaxel; Abraxane
Drug: Ipilimumab — 3 mg/kg by vein over 90 minutes on day 1. Ipilimumab dose repeated every 21 days for a total of 4 doses.
  Other Names: Yervoy; BMS-734016; MDX010
Behavioral: Phone Call — Every 2 months for 6 months, then every 3 months for up to 2 years, participant contacted by telephone. Each call should last about 5 minutes.

SUMMARY:
The goal of this clinical research study is to learn if the combination of ipilimumab and ABI-007 (abraxane) can help to control metastatic melanoma. The safety of this drug combination will also be studied.

Ipilimumab is designed to increase the immune system's ability to fight cancer.

Abraxane is designed to stop cancer cells from making new DNA (the genetic material of cells). This may stop the cancer cells from dividing into new cells.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive ABI-007 by vein over about 30 minutes on Days 1, 8, and 15 of each 28-day cycle. During the first 3 months that you receive abraxane, you will also receive ipilimumab. You will receive ipilimumab by vein over about 90 minutes. You will receive it 4 times, each time about 3 weeks apart.

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Tests:

Every week, blood (about 1 teaspoon) will be drawn for routine tests.

Before each cycle of abraxane:

* Your performance status will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for tests of the immune system (first 3 cycles only).
* You will be asked about any other drugs you may be taking and about any side effects you may be having.
* If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.

Every 8 weeks (+/- 7 days), you will have a chest x-ray and CT scans or MRI scans performed to check the status of the disease.

Length of Study:

You may receive ipilimumab for up to 3 months. You may continue taking abraxane for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

If you stop receiving the study drugs for any reason, you will have an End-of-Treatment Visit.

End-of-Treatment Visit:

Within 14 days after you stop study treatment, you will come into the clinic for the End-of-Treatment Visit. At this visit, the following tests will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any other drugs you may be taking and any side effects you may be having.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If the study doctor thinks it is in your best interest, you will have a CT scan or MRI scan to check for side effects.

Every 2 months for 6 months, then every 3 months for up to 2 years, you will also be contacted by telephone or during a routine clinic visit to see how you are doing. If you are called, each call should last about 5 minutes.

This is an investigational study. Ipilimumab is FDA approved and commercially available for the treatment of metastatic melanoma. abraxane is FDA approved and commercially available for the treatment of metastatic breast cancer. It is investigational to use abraxane, either alone or in combination with ipilimumab, for the treatment of metastatic melanoma.

Up to 64 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented diagnosis of advanced stage IV or unresectable stage III mucosal or cutaneous melanoma are eligible.
2. They must have recurrent melanoma with measurable or evaluable sites of disease, 1.0 cm or larger, in order to assess the response to treatment by the immune-related response criteria (irRC).
3. Patients should not have been previously treated with cytotoxic drugs and immunotherapeutic agents for unresectable Stage III or Stage IV disease. Prior Ipilimumab in metastatic setting is not allowed. Prior therapy may include one line of targeted therapy for metastatic disease ie BRAF or MEK inhibitor. At least 3 weeks should have passed since the last dose of prior adjuvant interferon therapy and prior targeted therapies, and all previous therapy related toxicities should have resolved before starting study treatment. Prior adjuvant interferon is permitted. Prior cytotoxic therapy in adjuvant or metastatic setting is not allowed. Prior Ipilimumab in adjuvant setting is not allowed. Prior adjuvant therapy with targeted therapy including but not limited to B-RAF, MEK inhibitors etc. is allowed. Prior palliative radiation therapy for metastatic melanoma is permitted provided the patient has unirradiated metastatic sites for response evaluation and has fully recovered from its toxicity.
4. Patients between 12 years of age and 70 years of age with an ECOG performance status of 0 or 1 will be eligible
5. They should have normal blood counts with a white blood cell count of more than or equal to 3000/mm^3 an absolute neutrophil count of more than or equal to 1500/mm^3 and a platelet count of more than 100,000/mm^3, Hemoglobin > 9.0 g/dL and have no impairment of renal function (serum creatinine less than 1.1 mg/dl for females and less than 1.4 mg/dl for males), hepatic function (serum bilirubin level of less than 1.5 mg/dl, AST and ALT </= 2.5X ULN unless presence of hepatic metastasis in which case AST and ALT </= 5X ULN are acceptable. Alk Phos </= 2.5X ULN ) and no evidence of significant cardiac or pulmonary dysfunction.
6. They should have no significant intercurrent illness such as an active infection associated with fever lasting more than 24 hours requiring antibiotics, uncontrolled psychiatric illness, hypercalcemia (calcium greater than 11 mg), or active GI bleeding. Females of child-bearing potential (non-childbearing is defined as greater than one year post-menopausal or surgically sterilized) must use acceptable contraceptive methods( abstinence, intrauterine device, oral contraceptive or double barrier devices) and must have a negative serum or urine pregnancy test within 72 hours prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study and signed informed consent .

Exclusion Criteria:

1. Patients with metastatic uveal melanoma
2. Patients with bone metastases only.
3. Patients with symptomatic brain or spinal cord metastases or requiring steroid therapy and patients with leptomeningeal disease. Patients with treated and stable CNS metastasis for 3 months or more, off steroids are eligible for the study. No major surgery or radiation therapy within 21 days before starting treatment.
4. Patients with significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricle function (Ejection Fraction less than 50%) on account of any organic disease such as hypertension or valvular heart disease or serious cardiac arrhythmia requiring therapy. Patients with significant history of cardiac disease will be evaluated by the investigator or his designee.
5. Patients with significant impairment of pulmonary function on account of chronic bronchitis, emphysema or chronic obstructive pulmonary disease (COPD) which has resulted in impairment of vital capacity of FEV1 to less than 75% of predicted normal values.
6. Patients with symptomatic effusions on account of pleural, pericardial or peritoneal metastases of melanoma.
7. Patients who are unable to return for follow-up visits as required by this study. Patients with a history of second malignant tumor, other than the common skin cancers - basal and squamous carcinomas, within the past 3 years and uncertainty about the histological nature of the metastatic lesions. Cases with other types of malignancies should be reviewed and decided by the PI of the study.
8. Patients with ≥ grade 2 sensory neuropathy at baseline.
9. Patients who have had major surgery or radiation therapy within 21 days of starting treatment.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adi Diab, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants signed the consent, 2 participants did not received treatment (1) withdrew prior treatment and (1) not eligible due to angiosarcoma (no melanoma).
Period: Overall Study
Arm/Group | ABI-007 + Ipilimumab
Started | 19
Completed | 18
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABI-007 + Ipilimumab
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival Response to Abraxane Plus Ipilimumab Therapy
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v 1.1) was used. Complete Response (CR)= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, no new lesions; Partial Response (PR)= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 50 months
Measure: Median (Full Range); unit: months
Groups:
- ABI-007 + Ipilimumab: Starting dose of ABI-007 is 150 mg/m2 administered by vein on days 1, 8, 15 every 28 days. Ipilimumab 3 mg/kg by vein over 90 minutes on day 1. Ipilimumab dose repeated every 21 days for a total of 4 doses.
Arm/Group | ABI-007 + Ipilimumab
Number analyzed (Participants) | 18
months | 24.9 [0 to 49]

2. Primary Outcome: Median Progression Free Survival
Description: Progression-free survival (PFS) is the time from random assignment in a clinical trial to disease progression or death from any cause.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABI-007 + Ipilimumab
Number analyzed (Participants) | 18
months | 10 [0.0 to 27.2]

ADVERSE EVENTS:
Time Frame: up to 50 months
Arm/Group | ABI-007 + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-007 + Ipilimumab (N=18)
Wound Infection (Investigations) | 1
Hypophysitis (Endocrine disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Cardiac disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Macular Cystoid (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-007 + Ipilimumab (N=18)
Alopecia (Skin and subcutaneous tissue disorders) | 18
Fatigue (General disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 16
Neuropathy (Nervous system disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Diarrhea (Gastrointestinal disorders) | 14
Pruritis (Skin and subcutaneous tissue disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Pain (General disorders) | 12
Anorexia (Metabolism and nutrition disorders) | 11
Nausea (Gastrointestinal disorders) | 11
Transaminitis (Investigations) | 11
Anemia (Blood and lymphatic system disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Headache (Nervous system disorders) | 7
Hypertension (Cardiac disorders) | 5
Chills (General disorders) | 4
Fever (General disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Mucositis (Gastrointestinal disorders) | 3
Elevated Bilirubin (Investigations) | 2
Elevated Creatinine (Investigations) | 2
Hypophysitis (Endocrine disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT01827111/Prot_SAP_000.pdf